CLINICAL TRIAL: NCT03518762
Title: Effect of Application of Sustained Lung Inflation on the Respiratory Outcome of Preterm Infants With Respiratory Distress Syndrome
Brief Title: Sustained Lung Inflation in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Douaa El Saied El Sherbiny, Doctor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 75381
Record Dates: First submitted 2018-04-12; First posted 2018-05-08 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained lung inflation (Experimental): Participants in this arm (n=80) received:
  1. Sustained lung inflation (SLI) manoeuvre(s) was applied once or twice, based on the protocol algorithm.
     Within the first 60 seconds of life, assessment for the need of advanced resuscitation (defined as the need for more than oxygen and tactile stimulation during resuscitation) was done;
     * Infants who needed advanced resuscitation were considered to receive SLI as a rescue approach.
     * Infants who needed only oxygen and tactile stimulation were considered to receive SLI as a prophylactic approach.
  2. Then Continuous positive airway pressure (CPAP). Intermittent positive pressure ventilation (IPPV) was given through an ETT, if intubation was needed.
  Interventions: Procedure: Sustained lung inflation (SLI); Procedure: Continuous positive airway pressure (CPAP)
- Control (Other): Participants in this arm (n=80) received:
  1. Resuscitation according to the American academy of pediatrics guidelines.
  2. Then Continuous positive airway pressure (CPAP). Intermittent positive pressure ventilation (IPPV) was given through an ETT, if intubation was needed.
  Interventions: Procedure: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Procedure: Sustained lung inflation (SLI) — SLI was given using a peak pressure of 20 cm H₂O sustained for 15 seconds,using a T-piece resuscitator, Neopuff device
  Arms: Sustained lung inflation
Procedure: Continuous positive airway pressure (CPAP) — CPAP through an appropriate mask using a pressure 5 cm H₂O,using a T-piece resuscitator, Neopuff device.

SUMMARY:
This is a randomized controlled study to investigate the effect of application of sustained lung inflation (SLI) at birth on the respiratory outcome of preterm infants with respiratory distress syndrome.

DETAILED DESCRIPTION:
Enrolled infants (n=160) were randomized before birth into 2 groups (intervention and control group) in a ratio 1:1. Randomization was done through an online randomizer (www.graphpad.com), and sealed envelopes were used to assign the infant to one of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 27 weeks and ≤ 32 weeks
* Appropriate for gestational age
* Weight >800 grams

Exclusion Criteria:

* Major congenital anomalies (congenital heart, cerebral, lung or abdominal malformations)
* Fetal hydrops

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2014-12-21 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Need for invasive mechanical ventilation or death | From birth up to 72 hours of life
  Treatment failure; defined as the need for intubation and invasive mechanical ventilation or death

SECONDARY OUTCOMES:
Duration of invasive mechanical ventilation | From date of birth until the date of discharge home or death from any cause, whichever came first, assessed upto 100 days
  The duration of intubation and invasive mechanical ventilation (in days)
Pneumothorax | From date of birth until the date of discharge home or death from any cause, whichever came first, assessed upto 100 days
  Pneumothorax, documented by radiological findings
Bronchopulmonary dysplasia | Assessed at 36 weeks postmenstrual age or discharge, whichever came first
  Bronchopulmonary dysplasia, defined as the need for more than 21% oxygen for at least 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abuel Hamd WA, El Sherbiny DE, El Houchi SZ, Iskandar IF, Akmal DM. Sustained Lung Inflation in Pre-term Infants at Birth: A Randomized Controlled Trial. J Trop Pediatr. 2021 Jan 29;67(1):fmaa097. doi: 10.1093/tropej/fmaa097. PMID 33254237